CLINICAL TRIAL: NCT04378153
Title: A Master Protocol to Test the Impact of Discontinuing Chronic Therapies in People With Cystic Fibrosis on Highly Effective CFTR Modulator Therapy (SIMPLIFY)
Brief Title: Impact of Discontinuing Chronic Therapies in People With Cystic Fibrosis on Highly Effective CFTR Modulator Therapy
Acronym: SIMPLIFY
Status: Completed | Type: Observational
Sponsor: Nicole Hamblett (Other)
Collaborators: Cystic Fibrosis Foundation (Other); Dartmouth-Hitchcock Medical Center (Other); University of Washington (Other)
Responsible Party: Sponsor-Investigator, Nicole Hamblett, Professor of Pediatrics, Division of Pulmonary and Sleep Medicine, University of Washington School of Medicine Adjunct Professor, Biostatistics, University of Washington School of Medicine Co-Executive Director, Cystic Fibrosis Therapeutics Development, Seattle Children's Hospital
Organization: Seattle Children's Hospital (Other)
Other Study IDs: SIMPLIFY-IP-19
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; CF; Withdrawal; Trikafta; hypertonic saline; dornase alfa; pulmozyme
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Master Study Run-in: Participants enrolled in the run-in phase of the master protocol.

SUMMARY:
Despite the increasingly common use of cystic fibrosis transmembrane conductance regulator (CFTR) modulator therapies in treating CF, it is still largely unknown whether or not other chronic therapies can be safely stopped. The SIMPLIFY study is being done to test whether or not it is safe to stop taking inhaled hypertonic saline or Pulmozyme® (dornase alfa) in those people that are also taking Trikafta™.

Trikafta (elexacaftor/tezacaftor/ivacaftor) is a combination CFTR modulator therapy that was approved by the Food and Drug Administration for people with CF who have at least one F508del mutation. The three drugs that make up Trikafta work together to allow many more chloride ions to move into and out of the cells, improving the balance of salt and water in the lungs. These changes result in better clearance of mucus from the lungs and improvements in lung function.

Inhaled hypertonic saline and Pulmozyme (dornase alfa) also improve clearance of mucus from the lungs to support lung function and have been available to people with CF for many years. Both therapies are considered to be relatively burdensome and it is not known whether either therapy can improve or maintain lung function above what is already gained through Trikafta use.

The goal of the SIMPLIFY study is to get information about whether or not it is safe to stop either inhaled hypertonic saline or Pulmozyme (dornase alfa) by testing if there is a change in lung function in subjects with cystic fibrosis (CF) who are assigned to stop their chronic medication (either hypertonic saline or Pulmozyme) as compared to those who are assigned to keep taking their medication while continuing to take Trikafta.

DETAILED DESCRIPTION:
SIMPLIFY-IP-19 is a master protocol is designed to evaluate the independent effects of discontinuing hypertonic saline or dornase alfa in people with cystic fibrosis (CF) age 12 and older currently taking the highly effective modulator elexacaftor/tezacaftor/ivacaftor (ETI). The hypertonic saline and dornase alfa sub studies are identical open label two-arm randomized non-inferiority trials consisting of a 2-week run-in period, randomization to continue or discontinue hypertonic saline or dornase alfa, followed by a 6-week study period. Subjects taking only hypertonic saline (HS) or dornase alfa at trial entry will be randomized 1:1 to either continue or discontinue the applicable therapy (i.e. HS or dornase alfa). Subjects taking both hypertonic saline and dornase alfa at study entry will be randomized to participate in either the hypertonic saline or dornase alfa and will be randomized (1:1) to continue or discontinue the applicable therapy (i.e. HS or dornase alfa). After completion of the first study, eligible subjects may subsequently enroll in the alternative study.

This clinicalrials.gov registration, NCT04378153, summarizes the 2-week run-in and adherence period prior to participant enrollment in either the Hypertonic Saline or Dornase Alfa sub studies.

Two additional clincialtrials.gov records document the sub study specific enrollment and outcome measures.

Hypertonic Saline Study Record

* NCT06350461
* Brief Title: Impact of Discontinuing Hypertonic Saline in People With CF on Highly Effective CFTR Modulators- A SIMPLIFY Sub-Study (SIMPLIFY-HS)

Dornase Alfa Study Record

* NCT06350474
* Brief Title: Impact of Discontinuing Dornase Alfa in People With CF on Highly Effective CFTR Modulator Therapy-A SIMPLIFY Sub-Study (SIMPLIFY-DN)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF.
* Age ≥ 12 years at the Screening Visit.
* Forced expiratory volume in 1 second (FEV1) ≥ 70 % predicted at the Screening Visit if < 18 years old, and ≥ 60 % predicted at Screening Visit if ≥ 18 years old.
* Clinically stable with no significant changes in health status within the 7 days prior to and including the Screening Visit.
* Current treatment with elexacaftor/tezacaftor/ivacaftor (ETI) for at least the 90 days prior to and including the Screening Visit and willing to continue daily use for the duration of the study.
* Currently taking hypertonic saline (at least 3%) and/or dornase alfa for at least the 90 days prior to and including the Screening Visit and willing to continue daily use for the 2-week screening period.

Exclusion Criteria:

* Active smoking or vaping.
* Use of an investigational drug within 28 days prior to and including the Screening Visit.
* Changes to chronic therapy (e.g., ibuprofen, azithromycin, inhaled tobramycin, aztreonam lysine) within 28 days prior to and including the Screening Visit. This includes new airway clearance routines.
* Acute use of antibiotics (oral, inhaled or IV) or acute use of systemic corticosteroids for respiratory tract symptoms within 7 days prior to and including the Screening Visit.
* Chronic use of systemic corticosteroids at a dose equivalent to ≥ 10mg per day of prednisone within 28 days prior to and including the Screening Visit.
* Antibiotic treatment for nontuberculous mycobacteria (NTM) within 28 days prior to and including the Screening Visit.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with Cystic Fibrosis using either hypertonic saline or dornase alfa chronically (see eligibility criteria).
Sampling Method: Non-Probability Sample
Enrollment: 987 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Mayer-Hamblett, PhD, Principal Investigator — University of Washington/Seattle Children's; Alex Gifford, MD, FCCP, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (80):
- United States (80):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Tucson Cystic Fibrosis Center, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - CHOC Children's Hospital, Orange, California
  - Stanford University Medical Center, Palo Alto, California
  - Rady Children's Hospital and Health Center at the University of California San Diego, San Diego, California
  - University of California, San Francisco - Adult Center, San Francisco, California
  - University of California, San Francisco - Peds Center, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Central Florida Pulmonary Group, Orlando, Florida
  - The Nemours Children's Clinic - Orlando, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Saint Luke's Cystic Fibrosis Center of Idaho, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Tulane University, Metairie, Louisiana
  - Maine Medical Partners Pediatric Specialty Care, Portland, Maine
  - John Hopkins Hospital, Baltimore, Maryland
  - Boston Children's Hospital, Brigham & Women's Hospital, Boston, Massachusetts
  - University of Michigan, Michigan Medicine, Ann Arbor, Michigan
  - Wayne State University Harper University Hospital, Detroit, Michigan
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - The Minnesota Cystic Fibrosis Center, Minneapolis, Minnesota
  - Children's Mercy Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Billings Clinic, Billings, Montana
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Monmouth Medical Center, Eatontown, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Cohen Children's Medical Center of New York, Lake Success, New York
  - Beth Israel Medical Center, New York, New York
  - Columbia University Cystic Fibrosis Program, New York, New York
  - University of Rochester Medical Center Strong Memorial, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - New York Medical College at Westchester Medical Center, Valhalla, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital/University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cystic Fibrosis Program, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Hershey Medical Center Pennsylvania State University, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - University of Texas Southwestern / Children's Health, Dallas, Texas
  - University of Texas Southwestern, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - University of Texas Health Center at Tyler, Tyler, Texas
  - Primary Children's Cystic Fibrosis Center, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Providence Medical Group, Cystic Fibrosis Center, Spokane, Washington
  - West Virginia University - Morgantown, Morgantown, West Virginia
  - University of Wisconsin, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
  - Froedtert & Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gold LS, Hansen RN, Mayer-Hamblett N, Nichols DP, Gifford AH, Kloster M, Goss CH, Kessler L. The cost of simplifying treatments for cystic fibrosis: Implications of the SIMPLIFY trial. J Manag Care Spec Pharm. 2024 Jan;30(1):26-33. doi: 10.18553/jmcp.2024.30.1.26. PMID 38153868
- [Derived] Mayer-Hamblett N, Ratjen F, Russell R, Donaldson SH, Riekert KA, Sawicki GS, Odem-Davis K, Young JK, Rosenbluth D, Taylor-Cousar JL, Goss CH, Retsch-Bogart G, Clancy JP, Genatossio A, O'Sullivan BP, Berlinski A, Millard SL, Omlor G, Wyatt CA, Moffett K, Nichols DP, Gifford AH; SIMPLIFY Study Group. Discontinuation versus continuation of hypertonic saline or dornase alfa in modulator treated people with cystic fibrosis (SIMPLIFY): results from two parallel, multicentre, open-label, randomised, controlled, non-inferiority trials. Lancet Respir Med. 2023 Apr;11(4):329-340. doi: 10.1016/S2213-2600(22)00434-9. Epub 2022 Nov 4. PMID 36343646
- [Derived] Yang C, Montgomery M. Dornase alfa for cystic fibrosis. Cochrane Database Syst Rev. 2021 Mar 18;3(3):CD001127. doi: 10.1002/14651858.CD001127.pub5. PMID 33735508
- [Derived] Mayer-Hamblett N, Nichols DP, Odem-Davis K, Riekert KA, Sawicki GS, Donaldson SH, Ratjen F, Konstan MW, Simon N, Rosenbluth DB, Retsch-Bogart G, Clancy JP, VanDalfsen JM, Buckingham R, Gifford AH. Evaluating the Impact of Stopping Chronic Therapies after Modulator Drug Therapy in Cystic Fibrosis: The SIMPLIFY Clinical Trial Study Design. Ann Am Thorac Soc. 2021 Aug;18(8):1397-1405. doi: 10.1513/AnnalsATS.202010-1336SD. PMID 33465316

RESULTS

PARTICIPANT FLOW:
Groups:
- Master Study Run-in: These numbers represent the number of participants enrolled in the 2 week run-in period to be enrolled in a SIMPLIFY sub study.
  Individual Sub Study Enrollment can be found in:
  Hypertonic Saline Study Record
  * NCT06350461
  * Brief Title: Impact of Discontinuing Hypertonic Saline in People With CF on Highly Effective CFTR Modulators- A SIMPLIFY Sub-Study (SIMPLIFY-HS) Dornase Alfa Study Record
  * NCT06350474
  * Brief Title: Impact of Discontinuing Dornase Alfa in People With CF on Highly Effective CFTR Modulator Therapy-A SIMPLIFY Sub-Study (SIMPLIFY-DN)
Period: Overall Study
Arm/Group | Master Study Run-in
Started | 987
Completed | 903
Not Completed | 84

BASELINE CHARACTERISTICS:
Arm/Group | Master Study Run-in
Number analyzed (Participants) | 987
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.1 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 480
  Male | 507
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 67
  Not Hispanic or Latino | 920
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 950
  Race: Black or African American | 12
  Race: Asian | 2
  Race: American Indian or Alaskan Native | 1
  Race: Native Hawaiian or Other Pacific Islander | 0
  Race: Other, More than One Race, or Unknown/Not Reported | 22
FEV1 (% Predicted) [Mean (Standard Deviation); unit: Percent Predicted] — FEV1 % predicted is calculated using the Global Lung Initiative multi-ethnic reference equations for ages 3-95.
  Percent Predicted | 96.7 (16.8)
Current Medication Use [Count of Participants; unit: Participants]
  Dornase Alfa Only | 232
  Hypertonic Saline Only | 65
  Both Hypertonic Saline and Dornase Alfa | 690

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Eligible to be Assessed for Sub-study Enrollment
Description: The number of participants completing the run-in period of the study and not meeting any of the exclusion criteria during the run-in period.
Time Frame: 2-week run-in period
Measure: Count of Participants; unit: Participants
Arm/Group | Master Study Run-in
Number analyzed (Participants) | 987
Participants | 870
Statistical Analysis 1: Comparison: Master Study Run-in; Null hypothesis: proportion of participants changing assigned regimen is the same in Discontinue and Continue arms; Test type: Superiority; p = 0.1215, Fisher Exact; Difference in % Participants = 2.17, 95% CI 2-sided [-0.7 to 5.7] — Confidence interval calculated using the Newcombe-Wilson method without continuity correction. Direction of difference is Discontinue - Continue

ADVERSE EVENTS:
Time Frame: Adverse events were not collected during the run-in phase of the study.
Description: Adverse events were not collected during the run-in phase of the study.
Arm/Group | Master Study Run-in
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Adverse events were not collected as part of the run-in phase of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-02-14): https://cdn.clinicaltrials.gov/large-docs/53/NCT04378153/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-06): https://cdn.clinicaltrials.gov/large-docs/53/NCT04378153/SAP_001.pdf